CLINICAL TRIAL: NCT01162330
Title: The Benefits Feasibility and Acceptability of Extended Screening Testing in Newborn Babies Who Are Referred for Further Hearing Assessment After Their Neonatal Screen (BEST)
Brief Title: The Benefits Feasibility and Acceptability of Extended Screening Testing in Newborn Babies Who Are Referred for Further Hearing Assessment
Acronym: BEST
Status: Completed | Type: Observational
Sponsor: Newcastle-upon-Tyne Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 5286; 10/H0904/25 (Other: REC)
Record Dates: First submitted 2010-07-13; First posted 2010-07-14 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Hearing Loss; Cytomegalovirus
Keywords: Screening; Congenital Cytomegalovirus; CMV; Hearing loss
MeSH Terms: conditions — Hearing Loss; Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Babies referred for further hearing tests: Babies referred for further hearing tests after their neonatal hearing screening tests
  Interventions: Other: Screening urine and saliva tests for congenital Cytomegalovirus

INTERVENTIONS:
Other: Screening urine and saliva tests for congenital Cytomegalovirus — With consent for the study babies who are referred for further hearing tests will have a urine and saliva sample sent to be analysed for CMV infection

SUMMARY:
This study will look at the feasibility and acceptability of testing newborn babies who are referred after their newborn hearing screen for an infection called congenital Cytomegalovirus (cCMV). Around 1 in every 100 to 200 babies is born with this virus, and although most remain well it causes 1 in 5 cases of childhood deafness. Knowing that a baby is infected shortly after birth could have significant benefit since a treatment is now available, but screening programs need to be feasible and acceptable. This study aims to evaluate targeted screening for cCMV by taking samples (saliva and urine) from babies who do not pass their newborn hearing screening. The investigators want to see if we can find a quick, reliable and parentally acceptable way to screen babies who fail their hearing test for this virus.

ELIGIBILITY:
Inclusion Criteria:

* All infants 'referred' for one or both ears following hospital-based newborn hearing screening in North of Tyne and South West London areas. Babies with other known causes of SNHL (e.g. hereditary) and those admitted to Neonatal Intensive Care Units will be included.

Exclusion Criteria:

* Exclusions to this study will be infants with parents/guardians not willing/able to give informed consent or children known to have congenital CMV by antenatal testing or clinical features of CMV infection at birth.

Max Age: 21 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This population this study examines is infants in Newcastle and South West London who are referred for more hearing tests after their neonatal hearing screen.
  This cohort of patients will be offered screening tests for congenital CMV infection.
Sampling Method: Non-Probability Sample
Enrollment: 411 (Actual)
Dates: Start 2010-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Feasibility of targeted screening for congenital CMV | 30 months
  Feasibility: as determined by proportion of urine and salivary swabs processed with a result back to parents and health professionals that would allow treatment if needed to be initiated by 28 days of age.
Acceptability of extended screening tests | 30 months
  Parental acceptability as determined by anxiety measures (in comparison to published data in parents whose infants are referred for failing their hearing screen, but where no mention of extended screening is made) and parental responses to extended questionnaires about the ease of the process of obtaining samples.

SECONDARY OUTCOMES:
Clinical utility of extended screening tests | 30 months
  Secondary outcomes.
  Assess and compare the clinical utility of performing salivary and urine CMV testing on babies referred through NHSP in terms of:
  1. rate of diagnosis of cCMV by day 21
  2. rate of initiation of treatment, where clinically indicated, by 4 weeks of age. 2. Calculate the prevalence of cCMV in children with SNHL detected following newborn hearing screening (number per population screened)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Clark, Study Chair — Newcastle-upon-Tyne Hospitals NHS Trust; Janet Berrington, Principal Investigator — Newcastle-upon-Tyne Hospitals NHS Trust; Mike Sharland, Principal Investigator — St Georges Healthcare Trust; Suzanne Luck, Principal Investigator — Royal Free Hospital NHS Foundation Trust
Locations (1):
- Royal Victoria Infirmary, Newcastle Hospital NHS Trust, Newcastle upon Tyne, Tyne and Wear, United Kingdom